CLINICAL TRIAL: NCT03356223
Title: A Phase II Trial Aiming to Evaluate the Clinical Interest of ABEMACICLIB Monotherapy in Patients With Locally Advanced/Metastatic Head and Neck Cancer After Failure of Platinum and Cetuximab or Anti-EGFR-based Therapy and Harboring an Homozygous Deletion of CDKN2A, and/or an Amplification of CCND1 and/or of CDK6
Brief Title: Evaluation of ABEMACICLIB Monotherapy in Patients With Locally Advanced/Metastatic Head and Neck Cancer After Failure of Platinum and Cetuximab or Anti-EGFR-based Therapy and Harboring an Homozygous Deletion of CDKN2A, and/or an Amplification of CCND1 and/or of CDK6
Acronym: ABORL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET16-116 (ABORL)
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Cancer; Advanced Cancer; Metastatic Cancer
Keywords: Clinical Trial; Phase II; Monotherapy; Abemaciclib; Homozygous deletion of CDKN2A; Amplification of CCND1; Amplification of CDK6; Multicenter Trial
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abemaciclib (Experimental)
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — 400mg/day with 2 doses of 200mg 12-hour apart For each 28-day cycle, a total of 56 doses of study drug will be dispensed.
  Route of administration : oral
  Duration of treatment until the patient experiences an unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.

SUMMARY:
This trial is an open-label, single arm, Phase II study using an A'Hern single stage design.

The molecular prescreening step will allow to defined HPV tumor status as well as molecular status CDKN2A, CCND1 and CDK6. Following this centralized molecular screening, only patients with HPV negative status and with tumor harboring CDKN2A homozygous deletion and/or CCND1 amplification and/or CDK6 amplification could initiate abemaciclib at time of documented radiological progression. Patients will be treated with ABEMACICLIB, 400 mg/day with 2 doses of 200 mg 12 hour apart (QH12). A cycle is defined as an interval of 28 days. For each 28-day cycle, a total of 56 doses of study drug will be dispensed.

DETAILED DESCRIPTION:
SAMPLE SIZE DETERMINATION The primary endpoint is the non-progression rate (CR, PR, SD as per RECIST 1.1) after 8 weeks of treatment.

The sample size calculation was based on an A'Hern single stage phase II design, with a minimum success (non- progression) rate considered of interest of p1=40% and an uninteresting rate of p0=15%. Assuming a type I error alpha of 0.05 and 85% power, 23 patients are needed to reject the null hypothesis H0: p<=p0 vs the alternative hypothesis H1: p ≥ p1 in a unilateral situation.

Based on the assumption that 10% of the patients may be non-evaluable, 25 patients will be included in the study.

DATA ENTRY AND DATA MANAGEMENT All the data concerning the patients will be recorded in the eCRF throughout the study. SAE reporting will be paper-based by Fax.

The sponsor will perform the study monitoring and will help the investigators to conduct the study in compliance with the clinical trial protocol, Good Clinical Practices (GCP) and local low requirements.

ELIGIBILITY:
Inclusion Criteria:

* I1. Male or female patients aged ≥ 18 years at time of inform consent signature
* I2. Histologically proven metastatic or locally advanced HNSCC (oropharynx, oral cavity, hypopharynx and larynx). Patients with cancer of nasopharynx (i.e. cavum cancer) are not eligible
* I3. Availability of a representative formalin-fixed paraffin-embedded (FFPE) primary and/or metastatic tumor tissue with an associated pathology report for molecular pre-screening: either an archival tumor block or a dedicated freshly collected tumor biopsy.
* I4. Documented CDKN2A homozygous deletion and/or CCND1 amplification and/or CDK6 and/or CDK4 amplification and no deletion/losses more than single copy of RB1 by copy number data before C1D1.

Note: This molecular pre-screening will be centralized at at the CGH platform of Centre Léon Bérard (CLB).

Note: This molecular pre-screening will be centralized at the CGH platform of Centre Léon Bérard (CLB).

Note: This molecular pre-screening can be performed for patient without documented disease progression (PD) but study drug treatment cannot be initiated until confirmed radiological PD.

* I5. HPV negative tumor status must be documented before C1D1. Note: This analysis will be centralized and performed by translational Biopathology platform of CLB during molecular pre-screening by IHC for p16.
* I6. Documented radiological progression or relapse after at least platin and cetuximab or anti-EGFR-based chemotherapy (combination or sequential treatment) and other standard treatment available at time of C1D1..
* I7. At least one measurable lesion by CT-scan as per RECIST 1.1.
* I8. At least one biopsiable tumor lesion before C1D1 i.e. at least one lesion with a diameter of at least 10 mm, visible by medical imaging and accessible to percutaneous sampling.
* I9. Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1.
* I10. Life expectancy > 12 weeks.
* I11. Patients must be able to swallow capsules.
* I12. Adequate organ and bone marrow function as defined by the following tests (to be checked using medical records and then carried out within 7 days prior C1D1):

  * Bone marrow :

    * Absolute neutrophil count >= 1.0 x 109/L
    * Platelet count > 100 x 109/L
    * Hemoglobin value >= 9 g/dL Note : Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
  * Renal function

    * Calculated creatinine clearance by MDRD or CDK-EPI > 50mL/min/1.73m2
  * Liver function

    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (or < 5.0 x ULN if liver metastases are present)
    * Total serum bilirubin ≤ 1.5 x ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤ 3mg/dL is acceptable).
* I13. Women of childbearing potential (entering the study after a confirmed menstrual period and who have a negative pregnancy test within 7 days before C1D1) must agree to use two methods of medically acceptable forms of contraception from the date of negative pregnancy test up to 3 months after the last study drug intake.
* I14. Fertile males must use a highly effective contraception during dosing period and through 3 months after final dose of study drug.
* I15. Patient should be able and willing to comply with study visits and procedures as per protocol.
* I16. Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.
* I17. Patients must be covered by a medical insurance.

Exclusion Criteria:

* NI1. Cancer disease considered curable with surgery or radiotherapy.
* NI2. Patient with a concurrent malignancy or has a malignancy within 3 years of study enrollment (with the exception of adequately treated basal or squamous cell carcinoma or non-melanomatous skin cancer).
* NI3. Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of abemaciclib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* NI4. Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate her participation in the clinical study (for example, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis).
* NI5. Persisting significant toxicities related to prior treatments i.e. ≥ Grade 2 AE according to CTCAE V5.0 except alopecia (any grade), grade 2 peripheral neuropathy and biological values as defined in inclusion criteria.
* NI6. Hypersensitivity to the active substance or excipient of study drug.
* NI7. Have received prior treatment with any CDK4/6 inhibitor (or participated in any CDK4/6 inhibitor clinical trial for which treatment assignment is still blinded).
* NI8. Patient has received treatment with a drug that has not received regulatory approval for any indication within :

  * 14 days of C1D1 for non myelosuppressive agent or
  * 21 days of C1D1 for a myelosuppressive agent.
* NI9. Patient has had major surgery and/or radiotherapy within 14 days prior to C1D1.
* NI10. Patient has received within 28 days prior to C1D1 yellow fever vaccine.
* NI11. Patient has a personal history within the last 12 months prior to C1D1 of any of the following conditions: syncope of cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest.
* NI12. Patient needs for the following concomitant medications/interventions not permitted during the study treatment period:

  * Any investigational anticancer therapy other than the study drug.
  * Any concurrent chemotherapy, radiotherapy (except palliative radiotherapy after discussion with the Sponsor), immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
  * Major surgery.
  * Strong and moderate inducers and inhibitors of CYP3A (for example grapefruit or grapefruit juice, phenytoin and carbamazepine).
  * Enzyme-Inducing Anti-Epileptic Drugs (EIAED).
* NI13. Patient has received an autologous or allogeneic stem-cell transplant.
* NI14. Patient has an active systemic fungal and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies).
* NI15. Pregnant or breast-feeding female patients.
* NI16. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to C1D1and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days prior to C1D1. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
The 8-week non-progression rate defined as the rate of patients with complete response (CR), partial response (PR) or stable disease (SD) lasting at least 8 weeks, according to RECIST v1.1 | 8 weeks after start of treatment

SECONDARY OUTCOMES:
8-week Objective response rate | 8 weeks after start of treatment
  Objective response rate after 8 weeks is defined as the proportion of patients with complete or partial response after 8 weeks of treatment according to RECIST 1.1.
Duration of response | 12 months after start of treatment
  The Duration of Response (DoR) will be measured from the time of first documented response (CR or PR as per RECIST 1.1) until the first documented disease progression or death due to underlying cancer, or censored at the date of the last available tumor assessment
Best response rate | 12 months after start of treatment
Time to progression | 12 months after start of treatment
  The Time to Progression will be measured from the time of treatment start until the first documented disease progression
Time to Treatment failure | 12 months after start of treatment
  The Time to treatment failure will be measured from the time of treatment start until discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death
Progression Free survival | 12 months after start of treatment
  Progression-Free Survival (PFS) will be measured from the date of inclusion until the date of event defined as the first documented progression or death from any cause. Patients with no event at the time of the analysis will be censored at the date of the last available tumor assessment. PFS will be estimated using the Kaplan-Meier method
Overall Survival | 12 months after start of treatment
  Overall survival will be measured from the date of treatment start to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme FAYETTE, MD, Principal Investigator — Centre Leon Berard
Locations (3):
- France (3):
  - Hôpital Saint-André, Bordeaux
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lassagne, Nice

REFERENCES:
- [Background] Vokes EE, Weichselbaum RR, Lippman SM, Hong WK. Head and neck cancer. N Engl J Med. 1993 Jan 21;328(3):184-94. doi: 10.1056/NEJM199301213280306. No abstract available. PMID 8417385
- [Background] Molin Y, Fayette J. Current chemotherapies for recurrent/metastatic head and neck cancer. Anticancer Drugs. 2011 Aug;22(7):621-5. doi: 10.1097/CAD.0b013e3283421f7c. PMID 21131821
- [Background] Vermorken JB, Trigo J, Hitt R, Koralewski P, Diaz-Rubio E, Rolland F, Knecht R, Amellal N, Schueler A, Baselga J. Open-label, uncontrolled, multicenter phase II study to evaluate the efficacy and toxicity of cetuximab as a single agent in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck who failed to respond to platinum-based therapy. J Clin Oncol. 2007 Jun 1;25(16):2171-7. doi: 10.1200/JCO.2006.06.7447. PMID 17538161
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Fayette J, Montella A, Chabaud S, Bachelot T, Pommier P, Girodet D, Racadot S, Montbarbon X, Favier B, Zrounba P. Paclitaxel is effective in relapsed head and neck squamous cell carcinoma: a retrospective study of 66 patients at a single institution. Anticancer Drugs. 2010 Jun;21(5):553-8. doi: 10.1097/CAD.0b013e3283388e60. PMID 20220515
- [Background] Sherr CJ. Cancer cell cycles. Science. 1996 Dec 6;274(5293):1672-7. doi: 10.1126/science.274.5293.1672. PMID 8939849
- [Background] Ortega S, Malumbres M, Barbacid M. Cyclin D-dependent kinases, INK4 inhibitors and cancer. Biochim Biophys Acta. 2002 Mar 14;1602(1):73-87. doi: 10.1016/s0304-419x(02)00037-9. PMID 11960696
- [Background] Shapiro GI. Cyclin-dependent kinase pathways as targets for cancer treatment. J Clin Oncol. 2006 Apr 10;24(11):1770-83. doi: 10.1200/JCO.2005.03.7689. PMID 16603719
- [Background] Sherr CJ, Roberts JM. CDK inhibitors: positive and negative regulators of G1-phase progression. Genes Dev. 1999 Jun 15;13(12):1501-12. doi: 10.1101/gad.13.12.1501. No abstract available. PMID 10385618
- [Background] Michalides RJ, van Veelen NM, Kristel PM, Hart AA, Loftus BM, Hilgers FJ, Balm AJ. Overexpression of cyclin D1 indicates a poor prognosis in squamous cell carcinoma of the head and neck. Arch Otolaryngol Head Neck Surg. 1997 May;123(5):497-502. doi: 10.1001/archotol.1997.01900050045005. PMID 9158396
- [Background] Akervall JA, Michalides RJ, Mineta H, Balm A, Borg A, Dictor MR, Jin Y, Loftus B, Mertens F, Wennerberg JP. Amplification of cyclin D1 in squamous cell carcinoma of the head and neck and the prognostic value of chromosomal abnormalities and cyclin D1 overexpression. Cancer. 1997 Jan 15;79(2):380-9. PMID 9010112
- [Background] Liggett WH Jr, Sewell DA, Rocco J, Ahrendt SA, Koch W, Sidransky D. p16 and p16 beta are potent growth suppressors of head and neck squamous carcinoma cells in vitro. Cancer Res. 1996 Sep 15;56(18):4119-23. PMID 8797577
- [Background] Kothari V, Mulherkar R. Inhibition of cyclin D1 by shRNA is associated with enhanced sensitivity to conventional therapies for head and neck squamous cell carcinoma. Anticancer Res. 2012 Jan;32(1):121-8. PMID 22213296
- [Background] Chung CH, Zhang Q, Kong CS, Harris J, Fertig EJ, Harari PM, Wang D, Redmond KP, Shenouda G, Trotti A, Raben D, Gillison ML, Jordan RC, Le QT. p16 protein expression and human papillomavirus status as prognostic biomarkers of nonoropharyngeal head and neck squamous cell carcinoma. J Clin Oncol. 2014 Dec 10;32(35):3930-8. doi: 10.1200/JCO.2013.54.5228. Epub 2014 Sep 29. PMID 25267748